CLINICAL TRIAL: NCT04880421
Title: Diagnostic Performance of Arterial Time for CT Assessment of Parietal Enhancement Defect for the Diagnosis of Ischemia in Mechanical Small Bowel Occlusions: a Comparative Study With Portal Time
Acronym: PORTOGRELE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PORTOGRELE
Record Dates: First submitted 2021-04-26; First posted 2021-05-10 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Bowel Obstruction Small

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intestinal obstruction is a frequent cause of emergency room visits and represents about 4-7% of the causes of acute abdominal pain syndrome and up to 30% in adults over 60 years old.

Although 65 to 80% of patients are treated medically, small bowel obstruction remains a serious pathology, with a high mortality rate that can reach 25% in case of small bowel ischemia. It is necessary to systematically perform a CT scan in the initial workup of small bowel obstructions to confirm the diagnosis, identify the mechanism and detect signs of ischemia that would require emergency surgery.

The best sign for the diagnosis of ischemia is the defect or asymmetry of parietal enhancement of the dilated small bowel. In the literature, this sign is described almost exclusively at portal time. In case of suspicion of mesenteric ischemia (another serious pathology affecting the small bowel), it is recommended to perform an examination with three acquisitions (without injection, arterial time, and portal time).

The department's experience has shown that arterial time is sometimes more sensitive than portal time for visualizing a parietal enhancement defect of the small bowel in mechanical occlusions.

Very few studies have investigated the diagnostic performance of parietal enhancement asymmetry on arterial time in mechanical occlusions of the small bowel.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with a diagnosis of mechanical small bowel obstruction on CT performed between April 2014 and December 2019
* Patient who had a CT scan with at least 3 phases: injection-free, arterial time, portal time
* French-speaking patient

Exclusion Criteria:

* Patient who did not have surgery within the first 24 hours
* Patient with a history of abdomino-pelvic surgery in the month preceding the scan
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient who objects to the use of his or her data for this research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, over 18 years of age, with a diagnosis of mechanical small bowel obstruction on CT and having had a CT scan with at least 3 phases: injection-free, arterial time, portal time, were managed at GHPSJ between April 2014 and December 2019
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of arterial versus portal phase in CT for the evaluation of parietal enhancement defect | Year 1
  This ouctome corresponds to the evaluation of the sensitivity, specificity, positive predictive value and negative predictive value of the acquisition for parietal enhancement defect as a sign of ischemia.

SECONDARY OUTCOMES:
Inter-observer reproducibility of parietal enhancement defect analysis at arterial time | Year 1
  This outcome corresponds to the evaluation of the Kappa coefficient of inter-observer reproducibility.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Zins, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Zins M, Millet I, Taourel P. Adhesive Small Bowel Obstruction: Predictive Radiology to Improve Patient Management. Radiology. 2020 Sep;296(3):480-492. doi: 10.1148/radiol.2020192234. Epub 2020 Jul 21. PMID 32692296
- [Background] Millet I, Taourel P, Ruyer A, Molinari N. Value of CT findings to predict surgical ischemia in small bowel obstruction: A systematic review and meta-analysis. Eur Radiol. 2015 Jun;25(6):1823-35. doi: 10.1007/s00330-014-3440-2. Epub 2015 Apr 8. PMID 25850889
- [Background] Ohira G, Shuto K, Kono T, Tohma T, Gunji H, Narushima K, Imanishi S, Fujishiro T, Tochigi T, Hanaoka T, Miyauchi H, Hanari N, Matsubara H, Yanagawa N. Utility of arterial phase of dynamic CT for detection of intestinal ischemia associated with strangulation ileus. World J Radiol. 2012 Nov 28;4(11):450-4. doi: 10.4329/wjr.v4.i11.450. PMID 23251723
- [Background] Chuong AM, Corno L, Beaussier H, Boulay-Coletta I, Millet I, Hodel J, Taourel P, Chatellier G, Zins M. Assessment of Bowel Wall Enhancement for the Diagnosis of Intestinal Ischemia in Patients with Small Bowel Obstruction: Value of Adding Unenhanced CT to Contrast-enhanced CT. Radiology. 2016 Jul;280(1):98-107. doi: 10.1148/radiol.2016151029. Epub 2016 Feb 11. PMID 26866378